CLINICAL TRIAL: NCT05453955
Title: Influence of Propofol and Remimazolam on Intraoperative Responses of Motor Evoked Potentials During Spine Surgery
Brief Title: Effect of Remimazolam on Motor Evoked Potential
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Seok Kyeong Oh, Assistant Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2022GR0051
Record Dates: First submitted 2022-07-08; First posted 2022-07-12 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol-Remimazolam (Experimental): General anesthesia was induced and maintained with propofol, then switched to remimazolam after 60 minutes from incision.
  Interventions: Drug: Propofol; Drug: Remimazolam Besylate
- Remimazolam-Propofol (Experimental): General anesthesia was induced and maintained with remimazolam, then changed to propofol after 60 minutes from incision.
  Interventions: Drug: Propofol; Drug: Remimazolam Besylate

INTERVENTIONS:
Drug: Propofol — Anesthesia induction and maintenance with propofol 60 minutes later, change the maintenance drug to remimazolam
  Other Names: Remimazolam Besylate
Drug: Remimazolam Besylate — Anesthesia induction and maintenance with remimazolam 60 minutes later, change the maintenance drug to propofol
  Other Names: Propofol

SUMMARY:
This study was planned to investigate the degree of effect of remimazolam on MEP compared to propofol when monitoring the motion-inducing potential (MEP).

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-70
* Scheduled for elective spine surgery requiring monitoring of evoked potential
* ASA physical status 1-3

Exclusion Criteria:

* BMI ≥ 40
* Uncontrolled DM (HbA1c ≥ 9%)
* Contraindications to the study drug: known allergy or hypersensitivity
* Use of rate responsive cardiac pacemaker with bioelectrical impedence
* Diagnosed neuromuscular disorder
* Pre-existing motor weakness

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-07 (Actual)

PRIMARY OUTCOMES:
Motor evoked potential (MEP), before cross-over | Intraoperative, just after confirmation of neuromuscular recovery, for 30 minutes
  Amplitude and latency of MEP before cross-over
MEP, after cross-over | Intraoperative, 30 minutes after alteration of the maintenance drug, for 30 minutes
  Amplitude and latency of MEP after cross-over

SECONDARY OUTCOMES:
Bispectral index | Intraoperative
  Bispectral index during MEP data collection
Blood pressure | Intraoperative
  Blood pressure during MEP data collection
Heart rate | Intraoperative
  Heart rate during MEP data collection

CONTACTS AND LOCATIONS:
Overall Officials: Sang Sik Choi, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Seok Kyeong Oh, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No